CLINICAL TRIAL: NCT00278252
Title: Phase II Study of Intravenous Etoposide in Patients With Relapsed Ependymoma
Brief Title: Etoposide in Treating Young Patients With Relapsed Ependymoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-CNS-2001-4; CDR0000454543 (Registry Identifier: PDQ (Physician Data Query)); EU-20576
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood ependymoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Familial ependymoma | interventions — Etoposide

INTERVENTIONS:
Drug: etoposide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well etoposide works in treating young patients with ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in young patients with relapsing and/or refractory ependymoma treated with a rapid schedule of intravenous etoposide.

Secondary

* Determine the possibility of second surgery or additional radiotherapy in these patients.

OUTLINE: This is a multicenter study.

Patients receive etoposide IV over 1 hour on days 1-3, 8-10, and 15-17. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients whose tumor becomes resectable after courses 3 or 6 undergo surgical resection.

After completion of study treatment, patients are followed periodically for approximately 5 years.

PROJECTED ACCRUAL: At least 14 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial ependymoma at first, second, or third relapse

  * Anaplastic (malignant) or low-grade ependymoma (cellular, papillary, clear cell, or mixed variants)
* Unequivocal evidence of tumor recurrence or progression by MRI scan after failing conventional treatment (e.g., primary surgery and adjuvant radiotherapy) for initial or recurrent disease
* Unresectable disease OR not amenable to complete surgical resection
* Measurable enhancing or non-enhancing disease on baseline scan performed within the past 2 weeks

  * Patients who have undergone prior surgery must have residual measurable disease

PATIENT CHARACTERISTICS:

* Lansky performance status 30-100%
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Serum total bilirubin normal
* AST < 2 times upper limit of normal
* No unrelated medical condition (e.g., renal or liver impairment) that would preclude chemotherapy treatment
* No active infection
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No radiotherapy within the past 6 weeks
* No chemotherapy within the past 4 weeks
* Prior IV etoposide allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2001-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Response rate by MRI after course 3

SECONDARY OUTCOMES:
Second surgery or additional radiotherapy in responding patients as assessed by MRI scan after course 3 or 6

CONTACTS AND LOCATIONS:
Overall Officials: Linda S. Lashford — The Christie NHS Foundation Trust; Susan V. Picton, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom

REFERENCES:
- [Derived] Apps JR, Maycock S, Ellison DW, Jaspan T, Ritzmann TA, Macarthur D, Mallucci C, Wheatley K, Veal GJ, Grundy RG, Picton S. Phase II study of intravenous etoposide in patients with relapsed ependymoma (CNS 2001 04). Neurooncol Adv. 2022 Apr 13;4(1):vdac053. doi: 10.1093/noajnl/vdac053. eCollection 2022 Jan-Dec. PMID 35591977